CLINICAL TRIAL: NCT05222295
Title: Comparison of the Effectiveness of Supervized Home-Based Pulmonary Telerehabilitation Program and Cognitive Telerehabilitation in Patients With Severe Chronic Obstructive Pulmonary Disease
Brief Title: The Effectiveness Pulmonary Telerehabilitation and Cognitive Telerehabilitation in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Amine Ataç, MSc Physiotherapist, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PulmoCogniRehab
Record Dates: First submitted 2022-01-22; First posted 2022-02-03 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Severe Chronic Obstructive Pulmonary Disease; Dyspnea; Muscle Weakness; Fatigue; Quality of Life; Muscle Strength; Motor Imagery; Functional Capacity; Muscle; Accessory; Respiratory Disease; Pulmonary Disease; COPD
Keywords: severe COPD; Severe Chronic Obstructive Pulmonary Disease; Pulmonary Telerehabilitation; Cognitive Telerehabilitation; Motor Imagery; Action Observation; Dyspnea; Muscle Strength; Blood Lactate Level; Daily Living Activities; Quality of Life; Muscle Weakness; Functional Capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Muscle Weakness; Fatigue; Respiration Disorders; Lung Diseases

STUDY DESIGN:
Intervention Model Description: Randomized prospective clinical trial
Who Masked: Participant
Masking Description: Each patient will be interviewed and evaluated alone, and it will be ensured that they do not coincide with other patients who may be included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Pulmonary Telerehabilitation Group (Experimental): Three times a week for 8 weeks, a supervised and standardized pulmonary rehabilitation program will be applied in the form of telerehabilitation with simultaneous video conference method, accompanied by a specialist physiotherapist, while the patients are at home.
  Interventions: Other: Supervised Pulmonary Telerehabilitation
- Cognitive Telerehabilitation Group (Experimental): Motor imagery + action observation methods will be applied. In therapy, a video recording of each exercise in the supervised telerehabilitation group will be sent to the patients by the physiotherapist in accordance with the number of repetitions. At the end of the session, the cognitive telerehabilitation group will be asked to actively do the breathing exercises and active breathing techniques cycle in the supervised telerehabilitation group as well as to imagine with the instructions in the video recording, and commands will be given accordingly.
  Interventions: Other: Cognitive Telerehabilitation

INTERVENTIONS:
Other: Supervised Pulmonary Telerehabilitation — For pulmonary rehabilitation to be applied in the simultaneous telerehabilitation method, digital blood pressure measurement device, digital finger pulse oximeter device will be given to severe COPD patients for safe exercise and they will be informed about confidence intervals and how to use saturation and heart rate monitors. The relevant program and points to be considered will be delivered to the patients in the form of an online PDF brochure.
  Arms: Supervised Pulmonary Telerehabilitation Group
Other: Cognitive Telerehabilitation — These patients will be asked to do a standardized pulmonary telerehabilitation program three times a week for 8 weeks by watching videos consisting of commands and exercise videos transmitted to them, some of them by actively doing, imagining.
  Arms: Cognitive Telerehabilitation Group

SUMMARY:
The aim of our study is to compare the effectiveness of the supervized pulmonary telerehabilitation program and the cognitive telerehabilitation method, which includes pulmonary telerehabilitation methods, in patients with severe stage COPD who have difficulty exercising heavily. The effects of pulmonary and cognitive rehabilitation on dyspnea, muscle strength, functional capacity, quality of life, anxiety and depression levels in this patient group will be examined.

The number of studies in the literature in which the pulmonary rehabilitation program was applied as telerehabilitation is insufficient. Considering that this patient group is not motivated and has difficulty in exercising, motor imagery and movement observation methods from cognitive rehabilitation methods may be alternative methods for these patients. Although these methods have been very popular in recent years in terms of researching and demonstrating their effectiveness in various patient groups in the literature, no study has been found in which the effects of these methods have been applied in pulmonary disease groups. This study aims to contribute to the serious gap in the literature on the application of pulmonary telerehabilitation and its effectiveness, and to be an original study by investigating the effectiveness of motor imagery and action observation, which are popular rehabilitation methods of recent years, in COPD patients in the pulmonary disease group for the first time.

DETAILED DESCRIPTION:
The demographic information of the participants who accepted to participate in the study by reading and signing the voluntary consent form will be questioned with the demographic data form to be created by the researchers. The patients' dyspnea status will be evaluated with the Modified Medical Research Council Dyspnea Scale, and their exercise capacity will be evaluated with the 6-minute walk test (6 MWT). Modified Borg Scale will be used to determine dyspnea and leg fatigue before and after 6MWT, and a digital sphygmomanometer will be used to measure blood pressure. Before, during and after the test, saturation and heart rate will be determined by finger pulse oximetry. Blood lactate levels will be determined with a portable lactate meter. An electronic hand dynamometer will be used to measure peripheral muscle strength. Activities of daily living will be assessed with the London Chest Activity of Daily Living Scale. Quality of life will be determined by The Saint George Respiratory Questionnaire, and anxiety and depression status will be determined by the Hospital Anxiety and Depression Scale. Muscle activities will be analyzed using a surface electromyographic (EMG) measuring device. The mental imagery abilities of the patients will be evaluated with the Kinesthetic and Visual Imagery Questionnaire-20 and the mental chronometry method.

Evaluations will be made by the responsible physiotherapist at the hospital before the program, at the end of the 4th week and at the end of the 8th week of the program. The permissions for the use of the questionnaires to be used were obtained from the authors, who made the validity and reliability in Turkish, via e-mail. Ethical approval of the study was obtained from the Ethics Committee of Istanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being diagnosed with C and D group COPD according to GOLD (Global iniative for chronic Obstructive Lung Disease) staging
* Not using an assistive device
* Using the same drugs for the last 4 weeks
* Permission to participate in the exercise for the patient from the responsible physician
* Getting a score of 24 or higher in the Standardized Mini Mental State Examination (MMDM)
* Absence of additional comorbid diseases of the orthopedic, neurological, cardiac system
* Having a score of 30 or higher on each of the Kinesthetic and Visual Imagery Questionnaire -20 (KGIA-20) visual imagery score and kinesthetic imagery score

Exclusion Criteria:

* Refusing to participate in the study
* Presence of respiratory system disease other than COPD
* Contraindication for moderate-intensity exercise (eg, unstable heart disease or stage 2 hypertension)
* Being an active smoker
* Patients who have had an acute exacerbation of COPD in the last 4 weeks
* Patients who have used oral corticosteroid drugs in the last 4 weeks
* Internet, computer, etc. patients who do not have technological equipment
* Patients who had a COPD exacerbation during the study protocol
* Participants who cannot understand verbal instructions and are visually impaired
* Having participated in another clinical trial within the last 30 days and currently that could affect the results of the trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
The exercise capacity | Change from baseline functional capacity at 8 weeks
  The exercise capacity will be evaluate by the 6 minute walking test (6MWT).The test was conducted in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines.
Perception of dyspnea | Change from baseline dyspnea level at 8 weeks
  The patients' dyspnea status will be evaluated with the Modified Medical Research Council Dyspnea Scale (mMRC Dyspnea Scale). he severity of dyspnea is rated on a scale of 0 to 4. "0" means no dyspnea perception, "4" means severe dyspnea perception.
Peripheral muscle strength | Change from baseline peripheral muscle strength at 8 weeks
  An electronic hand dynamometer will be used to measure peripheral muscle strength.

SECONDARY OUTCOMES:
Respiratory muscle activity | Change from baseline accessory respiratory muscle activity at 8 weeks
  Main and accessory respiratory muscle activity will be analyzed using an electromyographic (EMG) measuring device.
Kinesthetic and Visual Imagery Questionnaire-20 | Change from baseline imagery abilities level at 8 weeks
  Patients' mental imagery abilities will be assessed with the Kinesthetic and Visual Imagery Questionnaire-20. With the questionnaire, the intensity level of the imagery is recorded on a 5-point Likert scale (Visual imagery; 5= As clear as the original, 4: Quite clear, 3= Medium sharp, 2= Blurred, 1= No image) (Kinesthetic imagery; 5= As intense as if you were doing the movement) , 4 = Fairly intense, 3 = Moderately intense, 2 = Slightly intense, 1 = no sensation).
Mental chronometry method | Change from baseline imagery abilities between real time and imagery time level at 8 weeks
  Patients' mental imagery abilities will be assessed with mental chronometry method.
Blood Lactate Measurement | Change from baseline blood lactate level at 8 weeks
  Measurement will be made from the middle finger with a portable blood lactate meter.
the London Chest Activity of Daily Living Scale | Change from baseline activities of daily living at 8 weeks
  Activities of daily living (ADL) will be assessed with the London Chest Activity of Daily Living Scale. Each item is scored from 0 to 5, and higher scores indicate greater difficulty in performing the ADL.
The Saint George Respiratory Questionnaire (SGRQ) | Change from baseline quality of life at 8 weeks
  Quality of life will be determined by The Saint George Respiratory Questionnaire. Scores range from 0-100. A score of zero indicates normal and a score of 100 indicates maximum disability. In the SGRQ questionnaire, four units of treatment-related change are considered significant.
the Hospital Anxiety and Depression Scale | Change from baseline anxiety and depression status at 8 weeks
  Anxiety and depression status will be determined by the Hospital Anxiety and Depression Scale. The items in the scale are evaluated with a 4-point Likert scale and are based on a scoring system between 0-3. According to the scoring, 0-1 is considered as non-patient, 2 as borderline patients, and 2-3 as severely ill.

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hansen H, Bieler T, Beyer N, Godtfredsen N, Kallemose T, Frolich A. COPD online-rehabilitation versus conventional COPD rehabilitation - rationale and design for a multicenter randomized controlled trial study protocol (CORe trial). BMC Pulm Med. 2017 Nov 16;17(1):140. doi: 10.1186/s12890-017-0488-1. PMID 29145831
- [Background] Blampain J, Ott L, Delevoye-Turrell YN. Seeing action simulation as it unfolds: The implicit effects of action scenes on muscle contraction evidenced through the use of a grip-force sensor. Neuropsychologia. 2018 Jun;114:231-242. doi: 10.1016/j.neuropsychologia.2018.04.026. Epub 2018 Apr 27. PMID 29709583